## The Safety and Efficacy of the Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) for Laser Laryngeal Surgery

## **Statistical Analysis Plan**

NCT03086265

February 24, 2020

The planned sample size for the study was 40 patients (subsequently reduced to 20 due to logistical constraints), randomized 1:1 to receive one of 2 oxygen delivery systems, Transnasal Humidified Rapid- Insufflation Ventilatory Exchange (THRIVE), or endotracheal tube (standard of care.

Anesthesia, surgical, and patient recovery outcomes were summarized using descriptive statistics, with p-values calculated using a 2-sided t-test and Fisher Exact test.